CLINICAL TRIAL: NCT02433314
Title: An Open Label, Expanded Access Protocol to Evaluate the Efficacy and Safety of SAGE-547 Injection in the Treatment of Subjects With Super-Refractory Status Epilepticus
Brief Title: An Open Label, Expanded Access Protocol With SAGE-547 for Super-Refractory Status Epilepticus
Status: No longer available | Type: Expanded Access
Sponsor: Supernus Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 547-SSE-302
Record Dates: First submitted 2015-04-29; First posted 2015-05-04 (Estimated); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Super-Refractory Status Epilepticus
MeSH Terms: interventions — brexanolone

INTERVENTIONS:
Drug: SAGE-547

SUMMARY:
This is an open-label, expanded access protocol, designed to offer treatment with SAGE-547 to subjects in SRSE, and to evaluate the efficacy and safety of SAGE-547 administered as a continuous intravenous infusion to these subjects

ELIGIBILITY:
Inclusion Criteria:

* Subjects six (6) months of age and older
* Subjects who have:

  * Failed to respond to the administration of at least one first-line agent (e.g., benzodiazepine or other emergent initial AED treatment), according to the institution's standard of care, and;
  * Failed to respond to at least one second-line agent (e.g., phenytoin, fosphenytoin, valproate, phenobarbital, levetiracetam or other urgent control AEDs), according to the institution's standard of care, and;
  * Not previously been administered a third-line agent but have been admitted to an intensive care unit with the intent of administering at least one third-line agent for at least 24 hours; or who have previously failed zero, one or more wean attempts from third-line agents and are now on continuous intravenous infusions of one or more third-line agents and in an EEG burst or seizure suppression pattern; or who have previously failed one or more wean attempts from third-line agents and are now either not on at least one continuous infusion of a third-line agent or are on one or more continuous infusions of third-line agents but not in an EEG burst or seizure suppression pattern.

Exclusion Criteria:

* Subjects with SRSE due to anoxic/hypoxic encephalopathy with highly malignant/ malignant EEG features
* Children (subjects aged less than 18 years) with an encephalopathy due to an underlying progressive neurological disorder
* Subjects who have any of the following:

  1. a GFR low enough to warrant dialysis for whatever reason, but dialysis is not planned or non-continuous dialysis is planned;
  2. severe cardiogenic or vasodilatory shock requiring two or more pressors that is not related to third-line agent use;
  3. fulminant hepatic failure;
  4. no reasonable expectation of recovery or life-expectancy of less than 30 days.
* Subjects who are being administered more than three third-line agents concomitantly or in whom the qualifying wean cannot be completed per protocol

Min Age: 6 Months | Sex: All
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Henrikas Vaitkevicius, MD, Principal Investigator — Brigham and Women's Hospital

REFERENCES:
- See also: Related Info — http://www.sagerx.com